CLINICAL TRIAL: NCT02588898
Title: B-Vitamins and Polyneuropathy in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Rima Obeid, Prof. (apl.) Dr., Universität des Saarlandes
Other Study IDs: B-vitamins polyneuropathy
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Complications
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fasting blood samples (serum, whole blood and EDTA-plasma)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes: Patients (both men and women) with diagnosed type 2 Diabetes for at least 5 years. Blood collection and electrophysiological tests were performed.
  Interventions: Device: Blood collection and electrophysiological tests
- Controls free of diabetes: Controls (both men and women) are people of the same age who are free of Diabetes. Blood collection and electrophysiological tests were performed.
  Interventions: Device: Blood collection and electrophysiological tests

INTERVENTIONS:
Device: Blood collection and electrophysiological tests — Blood collected using a conventional method. Electrophysiology was tested after nerve Stimulation. Medical history and symptoms were collected after a standardized interview.

SUMMARY:
This case-control study investigated B-vitamin and homocysteine in relation to the presence or the absence of type 2 diabetes and clinical signs of polyneuropathy.

DETAILED DESCRIPTION:
Blood samples were collected and clinical investigations were performed at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with or without diabetes.

Exclusion Criteria:

* Usage of supplements containing B-vitamins, methotrexate treatment, cerebral or cardiac events in the last three months
* Liver or renal dysfunction.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female subjects with or without diabetes.
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Red blood cell cobalamin levels | Baseline
Polyneuropathy grade estimated using a score including a combination of data from questionnaire and electrophysiology investigations | Baseline
  Polyneuropathy grade was accessed using a questionnaire and a clinical examination (electrophysiology) after nerve stimulation. A score includes the combination of questionnaire data and electrophysiology data.

SECONDARY OUTCOMES:
Plasma methylmalonic acid levels | Baseline
Plasma choline levels | Baseline
Plasma cobalamin levels | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rima Obeid, Dr., Principal Investigator — University Hospital of the Saarland, Department of Clinical Chemistry
Locations (1):
- University of Saarland, Homburg, Saarland, Germany

REFERENCES:
- [Result] Obeid R, Jung J, Falk J, Herrmann W, Geisel J, Friesenhahn-Ochs B, Lammert F, Fassbender K, Kostopoulos P. Serum vitamin B12 not reflecting vitamin B12 status in patients with type 2 diabetes. Biochimie. 2013 May;95(5):1056-61. doi: 10.1016/j.biochi.2012.10.028. Epub 2012 Nov 17. PMID 23168250
- [Derived] Obeid R, Awwad HM, Rabagny Y, Graeber S, Herrmann W, Geisel J. Plasma trimethylamine N-oxide concentration is associated with choline, phospholipids, and methyl metabolism. Am J Clin Nutr. 2016 Mar;103(3):703-11. doi: 10.3945/ajcn.115.121269. Epub 2016 Feb 10. PMID 26864355